CLINICAL TRIAL: NCT04434729
Title: Fetal Treatment of Galenic Malformations
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Darren Orbach (Other)
Responsible Party: Sponsor-Investigator, Darren Orbach, Chief, Neurointerventional Radiology, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00034727; 2020P000216 (Other: Partners Healthcare IRB)
Record Dates: First submitted 2020-06-13; First posted 2020-06-17 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Vein of Galen Malformations
MeSH Terms: conditions — Vein of Galen Malformations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Fetal embolization of vein of Galen malformation (Experimental): This is a single-arm study. Fetal subjects will undergo a one-time intervention of fetal embolization of vein of Galen malformation.
  Interventions: Device: Fetal embolization of vein of Galen malformation using Target XL and XXL Detachable Coils

INTERVENTIONS:
Device: Fetal embolization of vein of Galen malformation using Target XL and XXL Detachable Coils — The study involves a single fetal intervention of maternal transuterine, fetal transcranial torcular puncture and median prosencephalic vein embolization. Detachable platinum coils (Target XL and XXL Detachable Coil, Stryker Neurovascular) will be used to pack the prosencephalic varix.

SUMMARY:
This is a prospective, single-arm non-randomized interventional study of fetuses to assess the safety and efficacy of fetal embolization of Vein of Galen Malformation (VOGM). Subjects will receive a one-time study intervention of fetal embolization. Follow-up assessments will be collected every 4 weeks until delivery, as per standard of care. After delivery, neurological assessments will be performed every 6 months for 2 years (adjusted for gestational age). Data will be compared to historical cohorts.

DETAILED DESCRIPTION:
The study involves a single fetal intervention of maternal transuterine, fetal transcranial torcular puncture and median prosencephalic vein embolization. Detachable platinum coils (Target XL and XXL Detachable Coil, Stryker Neurovascular) will be used to pack the prosencephalic varix. This procedure will take place in an obstetric OR at Brigham and Women's Hospital. Data will be collected every 4 weeks post-procedure until delivery, as per standard of care. Data regarding delivery and post-delivery status will also be collected until the subject is discharged from the hospital. After delivery, neurological assessments will be performed every 6 months for 2 years (adjusted for gestational age). Data will be compared to historical cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman carrying a fetus harboring a vein of Galen malformation in whom the straight sinus or falcine sinus draining the prosencephalic varix measures 7 mm or more on fetal MRI (medio-lateral diameter measured at the narrowest point of the sinus along the rostral-caudal axis, assessed on a T2-weighted coronal slice).
* Fetal gestational age between 23 weeks and term as determined by clinical information and evaluation of first ultrasound.
* Anatomic diagnosis of fetal vein of Galen malformation.
* Well preserved brain parenchyma.
* Maternal age of 18 years and older.
* Eligible for continuous lumbar epidural anesthesia.
* Able to travel to study site for study evaluation, procedures and visits.

Exclusion Criteria:

* Extensive fetal brain parenchymal injury/gliosis, >10% of supratentorial brain volume (i.e., SFP presentation). This is a degree of fetal brain injury beyond which the risk of significant neurological morbidity is high, based on studies of prenatal ischemic stroke.
* Irreversible fetal non-brain organ injury (e.g. hydrops fetalis as a manifestation of heart failure, a finding which portends fatal outcome in fetuses with vein of Galen malformation), i.e., SFP presentation.
* Fetus with VOGM in whom the straight sinus or falcine sinus draining the prosencephalic varix measures less than 7 mm on fetal MRI (T2-weighted coronal slice, medio-lateral diameter measured at the narrowest point of the sinus along the anterior-posterior axis), fitting fetal MRI criteria for likely evolution into the IT cohort.
* Severe maternal obesity pre-pregnancy as defined by body mass index (BMI) of 40 or greater.
* Fetuses with major congenital anomalies.
* Evidence of preterm labor, rupture of membranes or abruption.
* Maternal coagulopathy: INR > 1.2; PT/PTT above normal ranges for the lab; platelets <100.
* Medical disease requiring current anticoagulation including maternal deep vein thrombosis.
* Prior maternal medical history that would preclude epidural anesthesia.
* Multi-fetal pregnancy.
* Placenta previa or accreta.
* Participation in another fetal study that influences maternal and fetal morbidity and mortality.
* Known maternal hypersensitivity to 316LM stainless steel.
* Supine hypotensive syndrome.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2026-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Darren Orbach, MD PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Orbach DB, Shamshirsaz AA, Wilkins-Haug L, Guseh S, Krispin E, Tworetzky W, O'Leary B, Larson AM, Rangwala SD, Oushy S, See AP. In Utero Embolization for Fetal Vein of Galen Malformation. JAMA. 2025 Sep 9;334(10):878-885. doi: 10.1001/jama.2025.12363. PMID 40788723
- [Derived] Orbach DB, Wilkins-Haug LE, Benson CB, Tworetzky W, Rangwala SD, Guseh SH, Gately NK, Stout JN, Mizrahi-Arnaud A, See AP. Transuterine Ultrasound-Guided Fetal Embolization of Vein of Galen Malformation, Eliminating Postnatal Pathophysiology. Stroke. 2023 Jun;54(6):e231-e232. doi: 10.1161/STROKEAHA.123.043421. Epub 2023 May 4. No abstract available. PMID 37139817
- [Derived] See AP, Wilkins-Haug LE, Benson CB, Tworetzky W, Orbach DB. Percutaneous transuterine fetal cerebral embolisation to treat vein of Galen malformations at risk of urgent neonatal decompensation: study protocol for a clinical trial of safety and feasibility. BMJ Open. 2022 May 24;12(5):e058147. doi: 10.1136/bmjopen-2021-058147. PMID 35613814

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fetal Embolization of Vein of Galen Malformation
Started | 7
Completed | 5
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fetal Embolization of Vein of Galen Malformation
Number analyzed (Participants) | 7
Age, Continuous [Mean (Full Range); unit: years] | 32.4 [22 to 36]
Sex: Female, Male [Count of Participants; unit: Participants] — Fetal sex
  Participants
    Female | 3
    Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 1
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Prenatal Safety of Fetal Embolization for Patients With Vein of Galen Malformations
Description: The procedure is deemed safe if
  1. None of the following unacceptable events occur within 7 days of fetal embolization:
     1. Fetal death
     2. Fetal intracranial hemorrhage, either parenchymal or extra-axial, other than petechial hemorrhage.
     3. Maternal death
  2. None of the following unacceptable events occur between fetal embolization and delivery:
     1. Intra-procedural and post-procedural morbidity to the fetus and mother, probably related to the fetal intervention, e.g. placental abruption with subsequent sequelae
     2. Preterm delivery < 28 weeks, probably related to the fetal intervention
     3. Maternal blood transfusion or unanticipated surgical intervention, probably related to the fetal intervention
     4. Presence of fetal imaging evidence of new brain injury in a location or pattern unexpected for the natural history of vein of Galen malformation, probably related to the fetal intervention
Time Frame: From fetal embolization to delivery
Population: All 7 participants enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Fetal embolization of vein of Galen malformation
Number analyzed (Participants) | 7
Participants | 5

2. Secondary Outcome: Efficacy of Fetal Embolization for Patients With Vein of Galen Malformations
Description: The procedure is deemed efficacious if none of the following serious postnatal events occur within 30 days of birth:
  1. Urgent neonatal embolization is needed. Without fetal intervention, we'd expect 80% of the cohort to require such intervention.
  2. Neonatal death. Without fetal intervention, we'd expect a mortality rate of 40% in this cohort.
  3. Brain MRI within the first three weeks after birth reveals parenchymal brain injury (acute infarct or gliosis) affecting > 10% of the supratentorial brain volume. Without fetal intervention, we'd expect 30% of patients in this cohort to show this kind of injury.
Time Frame: Within 30 days of birth
Population: All participants who successfully completed the embolization procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Fetal embolization of vein of Galen malformation
Number analyzed (Participants) | 5
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of enrollment through 2 years post-delivery.
Description: The NCI-CTCAE v 5.0 system is used for maternal adverse events. The International Neonatal Consortium (INC) Neonatal Adverse Event Severity Scale is used for neonatal adverse events.
Arm/Group | Fetal Embolization of Vein of Galen Malformation
All-Cause Mortality (participants affected / at risk) | 3/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fetal Embolization of Vein of Galen Malformation (N=7)
Sinus tachycardia, hypotension (Cardiac disorders) | 1 (1)
Complete chorion-amnion separation (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fetal Embolization of Vein of Galen Malformation (N=7)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Preterm premature rupture of membranes (PPROM) (Pregnancy, puerperium and perinatal conditions) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT04434729/Prot_SAP_000.pdf